CLINICAL TRIAL: NCT06028906
Title: Research and Development of Innovative Method and Technology for Cerebral Perfusion Pressure Diagnosis
Brief Title: Research of Optimal Cerebral Perfusion Pressure Diagnosis
Acronym: optCPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Collaborators: Kaunas University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: OptCPP, ver B; MIP-20-216 (Other Grant/Funding Number: Research Council of Lithuania)
Record Dates: First submitted 2023-08-17; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Trauma, Brain; Hemorrhage Cerebral
Keywords: optimal cerebral perfusion pressure; optimal arterial pressure; cerebral autoregulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multimodal physiological monitoring and cerebral autoregulation monitoring — Patients are monitored routinely during their treatment in ICU. Multimodal physiological monitoring include continuous monitoring of arterial blood pressure (ABP), intracranial pressure (ICP) (if available), ETCO2 (if available), cerebral perfusion pressure (if available), cerebral blood flow velocity (CBFV) and ECG.
  Non-invasive cerebral autoregulation index Mx will by calculated as a Pearson correlation coefficient between slow ABP and slow CBFV waves.
  Invasive cerebral autoregulation index (Pressure reactivity index PRx) will by calculated as a Pearson correlation coefficient between slow ABP and slow ICP waves.
  Non invasive CBFV will be measured by using TCD device DWL Multi Dop-T. Invasive ICP will be measured by using Codman ICP Express or Raumedic ICP monitor.

SUMMARY:
The research will investigate the hypothesis that timely identification of the optimal value of the cerebral perfusion pressure (optCPP) or optimal arterial blood pressure (optABP) is possible after detecting informative episodes of arterial blood pressure (ABP) that reflects the physiological autoregulatory reactions of the cerebral blood flow,

This biomedical study will be conducted to test this hypothesis and to develop an algorithm for identification of optimal brain perfusion pressure within limited time (several tens of minutes).

The goal of this observational study is to test the method of timely optimal cerebral perfusion pressure value or optimal arterial pressure value in intensive care patients after brain surgery.

The main question it aims to answer are: how long it takes to identify optimal cerebral perfusion value when arterial blood pressure is changing within safe physiological limits.

Objectives of the study

1. To perform a prospective observational study by collecting multimodal physiological brain monitoring data: intracranial pressure (ICP), arterial blood pressure (ABP), End-tidal carbon dioxide (ETCO2), cerebral blood flow velocity (CBFV), ECG.
2. To perform a retrospective analysis of the accumulated clinical monitoring data, in order to create an algorithm for the identification of informative monitoring data fragments, according to which it would be possible to identify the optimal cerebral perfusion pressure (optCPP) value in a limited time interval (within a few or a dozen minutes).
3. To perform a retrospective analysis of accumulated clinical monitoring data, determining correlations of cerebral blood flow autoregulation and optCPP-related parameters with the clinical outcome of patients and with the risk of cerebral vasospasm or cerebral ischemia.

DETAILED DESCRIPTION:
Optimal cerebral perfusion pressure (optCPP) management requires at least 4 hours of patients' physiological data monitoring. Critical pathophysiological events in the injured brain happen in minutes, not in hours.

The research will investigate the hypothesis that timely identification of the optimal value of the cerebral perfusion pressure (optCPP) or optimal arterial blood pressure (optABP) is possible after detecting informative episodes of arterial blood pressure (ABP) that reflects the physiological autoregulatory reactions of the cerebral blood flow,

This biomedical study will be conducted to test this hypothesis and to develop an algorithm for identification of optimal brain perfusion pressure within limited time (several tens of minutes).

The goal of this observational study is to test the method of timely optimal cerebral perfusion pressure value or optimal arterial pressure value in intensive care patients after brain surgery.

The main question it aims to answer are: how long it takes to identify optimal cerebral perfusion value when arterial blood pressure is changing within safe physiological limits.

Objectives of the study

1. To perform a prospective observational study by collecting multimodal physiological brain monitoring data: intracranial pressure (ICP), arterial blood pressure (ABP), End-tidal carbon dioxide (ETCO2), cerebral blood flow velocity (CBFV), ECG.
2. To perform a retrospective analysis of the accumulated clinical monitoring data, in order to create an algorithm for the identification of informative monitoring data fragments, according to which it would be possible to identify the optimal cerebral perfusion pressure (optCPP) value in a limited time interval (within a few or a dozen minutes).
3. To perform a retrospective analysis of accumulated clinical monitoring data, determining correlations of cerebral blood flow autoregulation and optCPP-related parameters with the clinical outcome of patients and with the risk of cerebral vasospasm or cerebral ischemia.

Timely identification of optCPP value and diagnosis of cerebrovascular autoregulation (CA) will be performed according to the measured reaction of cerebral hemodynamics during the detected ABP(t) changes.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury patients
* Subarachnoid hemorrhage patients

Exclusion Criteria:

* persons with mental disorders, but who can give consent to participate in biomedical research;
* minors;
* students, if their participation in biomedical research is related to studies;
* persons living in care institutions;
* soldiers during their actual military service;
* employees of health care institutions where biomedical research is conducted, subordinate to the researcher;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients treated at Vilnius University Hospital Santaros Klinikos that undergo brain surgery after traumatic brain injury (TBI) or subarachnoid hemorrhage (SAH).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral autoregulation index (pressure reactivity index PRx) | PRx is measured when invasive intracranial pressure slow waves and arterial pressure slow waves are available during multimodal clinical data collection in ICU (up to 7 days).
  Negative values of cerebral autoregulation index (PRx<0) represent intact cerebral autoregulation, positive values (PRx>0) show impaired cerebral autoregulation.
Cerebral autoregulation index (mean flow index Mx) | Mx is measured when non-invasive cerebral blood flow slow waves and arterial pressure slow waves are available during multimodal clinical data collection in ICU (up to 7 days).
  Negative values of cerebral autoregulation index (Mx<0) represent intact cerebral autoregulation, positive values (Mx>0) show impaired cerebral autoregulation.
Optimal arterial blood pressure value | Optimal arterial blood pressure value is identified when PRx or Mx data are available during multimodal clinical data collection in ICU (up to 7 days).
  Optimal arterial blood pressure value is identified at the conditions of lowest values of cerebral autoregulation indexes by applying "U-shape" approximation on ABP and PRx (or Mx) data.
  Identified optimal arterial blood pressure value is assumed as a targeted arterial blood pressure value for personalized cerebral perfusion management in the cases when U-shape approximation is determined.

SECONDARY OUTCOMES:
Patients' outcome | GOS is evaluated at discharge from hospital and after 30 days of patient's hospital admission.
  Patients' outcome is evaluated according to Glasgow Outcome Score (GOS). GOS scores are: 1 - death, 2 - persistent vegetative state, 3 - severe disability, 4 - moderate disability, 5 - low disability.
Occurrence of cerebral ischemia and cerebral vasospasms | CT and CTA scans is performed routinely on 7th day after SAH or within period of 3-21 day after SAH if necessary.
  Occurrence of cerebral ischemia and cerebral vasospasms evaluated from Computed Tomography (CT) and Computed Tomography Angiography (CTA) scans

CONTACTS AND LOCATIONS:
Overall Officials: Saulius Rocka, Principal Investigator — Head of the Neurosurgery Center at Vilnius University Hospital Santaros klinikos
Locations (1):
- Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaleckas E, Putnynaite V, Lapinskiene I, Preiksaitis A, Serpytis M, Rocka S, Bartusis L, Petkus V, Ragauskas A. Impaired cerebral autoregulation detected in early prevasospasm period is associated with unfavorable outcome after spontaneous subarachnoid hemorrhage: an observational prospective pilot study. Ultrasound J. 2024 Apr 15;16(1):24. doi: 10.1186/s13089-024-00371-8. PMID 38619783